CLINICAL TRIAL: NCT03543839
Title: Pilot Trial of Belimumab in Early Lupus
Brief Title: Trial of Belimumab in Early Lupus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Cynthia Aranow, MD, Professor, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-0861
Record Dates: First submitted 2018-04-12; First posted 2018-06-01 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Erythematosus
Keywords: lupus; early lupus; belimumab; autoreactivity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: This is not a true cross-over study. Subjects are randomized to receive true drug or placebo in the initial phase and then those patients who were randomized to receive belimumab will be rerandomized to receive either study drug or placebo. Subjects randomized at baseline to receive placebo continue to receive placebo through the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug or placebo look identical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Belimumab (Active Comparator): Subjects in this arm will receive 200mg belimumab for self administration subcutaneously weekly for 2 years
  Interventions: Biological: Belimumab
- Belimumab/Placebo (Experimental): Subjects in this arm will receive 200mg belimumab for self administration subcutaneously weekly for 1 year and then placebo injections subcutaneously for 1 year.
  Interventions: Biological: Belimumab/Placebo
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo for self administration subcutaneously weekly for 2 years
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Belimumab — Subjects in this arm will receive 200mg belimumab subcutaneously weekly for 2 years
  Arms: Belimumab
Biological: Belimumab/Placebo — Subjects in this arm will receive weekly subcutaneous injections of 200mg belimumab for 1 year and then placebo subcutaneous injections for 1 year.
  Arms: Belimumab/Placebo
Other: Placebo — Subjects in this arm will receive weekly subcutaneous injections of placebo for 2 years
  Arms: Placebo

SUMMARY:
This two year study will evaluate the effects of giving belimumab (Benlysta) to patients with Early Lupus. Early lupus is a diagnosis of lupus within 2 years. Subjects will be randomized to receive belimumab or placebo during the first year. During the second year, subjects who were randomized to belimumab will be rerandomized to continue to receive belimumab or to receive placebo. The study will look at clinical effects as well as effects on the immune system.

DETAILED DESCRIPTION:
This protocol proposes that early treatment of Systemic Lupus Erythematous (SLE) may prevent tissue damage and may even lead to long-term remission of disease. This concept is supported by reports of SLE-associated autoimmunity that are detected serologically many years prior to any constitutional symptoms or specific tissue inflammation and immune dysregulation precedes the development of clinically apparent SLE. Belimumab (Benlysta) is an FDA approved medication and is a monoclonal antibody directed against B cell-activating factor (BAFF)/ B Lymphocyte Stimulator (BLyS). B cells maturing in environments with high BAFF levels are more likely to be autoreactive B cells. This is a double-blind placebo controlled trial of belimumab, in patients with early lupus, ie lupus diagnosed within 2 years. Thirty subjects will be randomized (2:1) to receive subcutaneous belimumab weekly or placebo. After a year of treatment, subjects receiving belimumab will be rerandomized (1:1) to receive belimumab or placebo. The primary outcome is B cell autoreactivity. Clinical efficacy including disease activity, flares, attainment of low disease activity or remission as well as surrogate cardiovascular biomarkers will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE per current ACR classification criteria
* Date of SLE diagnosis within 2 years of screening
* ANA positive (with a titer ≥ 80)
* anti-ds DNA antibody positive
* Mild to moderate disease activity define by a SLEDAI-2K ≥4
* Stable corticosteroid dose in the 4 weeks prior to screening ≤ 30mg/day.
* If on methotrexate, dose must be stable for 4 weeks
* Concomitant treatment with hydroxychloroquine unless documented inability to tolerate
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Negative serum pregnancy test (for women of child bearing potential)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for 16 weeks after completion of treatment

Exclusion Criteria:

* Previous exposure to disease modifying drugs such as azathioprine, mycophenolate mofetil, cyclophosphamide, or cyclosporine.
* Previous exposure to biologic therapies including rituximab, belimumab or other agents that have been investigated for SLE.
* Active renal or nervous system disease or disease activity fulfilling BILAG A criteria
* Use of high dose steroids (>0.5 mg/kg/ day) within the 4 weeks prior to screening
* Expectation (by the investigator) that the subject will require treatment with a disease modifying drug within the first 52 weeks of the study
* Hemoglobin: < 8.0 gm/dL
* Platelets: < 50,000/mm
* ANC < 1.0 x 103/mm
* AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
* Creatinine clearance ≤ 25ml/min per 1.73 m2
* Positive Hepatitis B or C serology (Hep B Surface antigen, Hep B core Ab or Hepatitis C antibody)
* History of positive HIV (HIV conducted during screening if applicable)
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 30 days prior to baseline or concurrently with belimumab
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies
* Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria)
* Hospitalization for treatment of infection within 60 days of Day 0.
* Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 0
* History of serious recurrent or chronic infection
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 365 days prior to Day 0
* Pregnancy (a negative serum pregnancy test must be obtained for all women of childbearing potential at screening; a urine pregnancy test must be negative < 7 days prior to first dose and monthly)
* Lactation
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of malignant neoplasm within the last 5 years with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk
* History of a primary immunodeficiency
* Have a significant IgG deficiency (IgG level < 400 mg/dL)
* Have an IgA deficiency (IgA level < 10 mg/dL)
* Have any other clinically significant abnormal laboratory value in the opinion of the investigator
* Comorbidities requiring corticosteroid therapy, including those which have required two or more courses of systemic courses of systemic corticosteroids within the previous 12 months
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of anergic autoreactive naïve B cells | Assessment at year 1
  The frequency of autoreactive B cells in the naïve subset will be identified by flow cytometry.

SECONDARY OUTCOMES:
Frequency of anergic autoreactive naïve B cells | Assessment at year 2
  The frequency of autoreactive B cells in the naïve subset will be identified by flow cytometry.
Frequency of autoreactivity in transitional B cells | Year 1
  The frequency of autoreactive B cells in the transitional B cell subset will be identified by flow cytometry.
Frequency of autoreactivity in transitional B cells | Year 2
  The frequency of autoreactive B cells in the transitional B cell subset will be identified by flow cytometry.
Time to reconstitution of B cell subsets in subjects in belimumab/placebo arm randomized to receive placebo after 1 year of belimumab therapy | Year 2
  B cell numbers decrease following belimumab; the time for B cell reconstituion will be determined
SRI (SLE Response Index) modified | Year 1
  Systemic lupus response index
SRI modified | Year 2
  Systemic lupus response index
Low lupus disease activity state (LLDAS) | Year 1
  LLDAS as defined by the Asia-Pacific Lupus Association
Low lupus disease activity state | Year 2
  LLDAS as defined by the Asia-Pacific Lupus Association
Remission | Year 1
  Remission defined by DORIS (Definition of Remission in SLE)
Remission | Year 2
  Remission defined by DORIS (Definition of Remission in SLE)
Flare of lupus disease | Through year 2
  Lupus flare will be measure using the SELENA-SLEDAI (Safety of Estrogens in Lupus Erythematosus National Assessment --Systemic Lupus Erythematosus Disease Activity Index) flare instrument or British Isles Lupus Assessment Group (BILAG) disease activity index
New Classification Criteria for SLE. | Through year 2
  Accumulation of new American College of Rheumatology (ACR) Classification criteria or Systemic Lupus International Cooperative Clinics (SLICC) criteria
Serologies | Through year 2
  Changes in titers of anti-DNA antibody levels
Complement levels | Through year 2
  Changes in measures of C3 and C4 (mg/dL)
Complement levels | Through year 2
  Changes in measures of C3, C4 (mg/dL)
Serum immunoglobulin levels | Through year 2
  Change from baseline of serum IgG, IgM and IgA (mg/dL)
Damage | Through year 2
  Damage accrual assessed using a SLE damage index
Cardiovascular biomarkers | Through year 2
  IgM phosphocholine antibody titers and proinflammatory HDL
Safety and tolerability (adverse events) | Through year 2
  All adverse events and serious adverse events will be collected
Frequency of autoreactivity in CD27+, IgD+ memory B cells | Year 1
  The frequency of autoreactive B cells in the CD27+, IgD+ B cell subset will be identified by flow cytometry.
Frequency of autoreactivity in CD27+, IgD+ memory B cells | Year 2
  The frequency of autoreactive B cells in the CD27+, IgD+ B cell subset will be identified by flow cytometry.
Frequency of autoreactivity in CD27+, IgD- B cells | Year 1
  The frequency of autoreactive B cells in the CD27+, IgD- B cell subset will be identified by flow cytometry.
Frequency of autoreactivity in CD27+, IgD- B cells | Year 2
  The frequency of autoreactive B cells in the CD27+, IgD- B cell subset will be identified by flow cytometry.
Frequency of autoreactivity in CD27-, IgD- B cells | Year 1
  The frequency of autoreactive B cells in the CD27-, IgD- B cell subset will be identified by flow cytometry.
Frequency of autoreactivity in CD27-, IgD- B cells | Year 2
  The frequency of autoreactive B cells in the CD27-, IgD- B cell subset will be identified by flow cytometry.
The absolute numbers of transitional B cells | Year 1
  The number of transitional B cells will be determined by flow cytometry.
The absolute numbers of transitional B cells | Year 2
  The number of transitional B cells will be determined by flow cytometry.
The absolute numbers of naïve B cells | Year 1
  The number of transitional B cells will be determined by flow cytometry.
The absolute numbers of naïve B cells | Year 2
  The number of naïve B cells will be determined by flow cytometry.
The absolute numbers of memory B cells | Year 1
  The number of memory B cells will be determined by flow cytometry.
The absolute numbers of memory B cells | Year 2
  The number of memory B cells will be determined by flow cytometry.
The absolute number of plasmablasts | Year 1
  The number of plasmablasts will be determined by flow cytometry.
The absolute number of plasmablasts | Year 2
  The number of plasmablasts will be determined by flow cytometry.
The absolute number of plasma cells | Year 1
  The number of plasma cells will be determined by flow cytometry.
The absolute number of plasma cells | Year 2
  The number of plasma cells will be determined by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, MD, Principal Investigator — Feinstein Institute for Medical Research, Northwell Health
Locations (1):
- Feinstein Institute, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided